CLINICAL TRIAL: NCT06929195
Title: Phase I Clinical Trial Evaluating the Tolerability, Pharmacokinetics, and Preliminary Efficacy of TQB2210 Injection in Subjects With Advanced Malignant Tumors
Brief Title: Clinical Trial to Evaluate the Tolerance of TQB2210 Injection
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2210-I-01
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2024-12

CONDITIONS: Advanced Malignant Tumours

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2210 Injection (Experimental): Dose escalation experiment:
  Intravenous infusion once of TQB2210 for injection every two weeks, 28 days as one treatment cycle.
  (1.0 mg/kg, 3.0 mg/kg, 8.0 mg/kg, 16.0 mg/kg, 24.0 mg/kg)
  Dose expansion experiment:
  Chose one or two appropriate dose groups in the dose escalation experiment to amplify.
  Interventions: Drug: TQB2210 Injection

INTERVENTIONS:
Drug: TQB2210 Injection — TQB2210 injection is a humanized monoclonal antibody against FGFR2b, which can bind to FGFR2b with high specificity. It inhibits tumor growth by blocking the signaling pathway mediated by fibroblast growth factor receptor. Its binding is concentration dependent.

SUMMARY:
TQB2210 injection is a humanized monoclonal antibody against FGFR2b, which can bind to FGFR2b with high specificity and inhibit tumor growth by blocking the signaling pathway mediated by fibroblast growth factor receptor. The aim of this experiment is to evaluate the tolerability, pharmacokinetics, and preliminary efficacy of TQB2210 injection in patients with advanced malignant tumors, and to assess its effectiveness and phase II recommended dose (RP2D) in advanced malignant tumors with FGFR2b overexpression, such as advanced gastric/gastroesophageal junction cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years old; Eastern Cooperative Oncology Group Performance Status (ECOG-PS), score: 0-1; The expected survival time is more than 3 months.
* At least one tumour lesion that can be evaluated according to Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 in the dose-escalation phase and at least one measurable lesion in the dose-expansion phase.
* Good function of major organs.
* Patients with advanced malignant tumours confirmed by histology or cytology, disease progression or intolerance after adequate standard treatment, lack of standard treatment options.
* Can provide tumor tissue specimens collected fresh or sliced within 6 months (preserved in wax blocks collected within 3 years) for further detection for FGFR2b expression
* Fertile subjects should agree that contraception must be used during the study and for 6 months after the end of the study; Women of childbearing age had a negative serum pregnancy test within 7 days prior to study enrollment and had to be non-lactating subjects.
* Evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Has had or is currently suffering from other malignant tumors
* There are diseases that affect intravenous injection and venous blood collection
* Adverse reactions from previous treatments have not recovered to CTCAE v5.0 Grade 1
* Received major surgical treatment, significant traumatic injury within 4 weeks prior to the first dose of TQB2210, or exist long-term unhealed wounds or fractures
* Subjects who experience any bleeding or bleeding events ≥ CTCAE grade 3 within 4 weeks prior to the first dose of TQB2210
* An arterial/venous thrombotic event occurred within 6 months prior to to the first dose of TQB2210
* Patients with active viral hepatitis that is poorly controlled
* Active syphilis patients requiring treatment
* A history of active pulmonary tuberculosis, idiopathic pulmonary fibrosis, institutional pneumonia, drug-induced pneumonitis/radiation pneumonia requiring treatment or active pneumonia with obvious clinical symptoms, interstitial pneumonia requiring treatment
* Subjects with any severe and/or uncontrolled illnesses
* Individuals who are preparing for or have previously undergone allogeneic bone marrow transplantation or solid organ transplantation
* History of hepatic encephalopathy
* Suffering from significant cardiovascular disease
* Active or uncontrolled severe infections
* Patients with renal failure requiring hemodialysis or peritoneal dialysis;
* Corneal defects, corneal ulcers, keratitis or keratoconus, history of corneal transplantation, or other known corneal abnormalities that may increase the risk of developing corneal ulcers within 6 months prior to the first treatment or currently present
* History of retinal disease or retinal detachment, or increased risk of retinal detachment according to the opinion of an ophthalmologist
* Acute ophthalmic diseases that continue to progress within the first 4 weeks of enrollment
* Unwilling to avoid using contact lenses during research treatment
* History of immunodeficiency, includingHuman Immunodeficiency Virus（HIV） positivity or other acquired or congenital immunodeficiency diseases
* There are poorly controlled autoimmune diseases that require the use of immunosuppressants or systemic hormone therapy to achieve immunity Subjects who inhibit the purpose and need to continue using it within 7 days before the first administration
* Individuals with epilepsy who require treatment
* Poor control of diabetes
* Tumor related symptoms and treatment:

  1. Received chemotherapy, immunotherapy, small molecule targeted drugs, etc. within 3 weeks before the first administration;
  2. Traditional Chinese patent medicines and simple preparations with anti-tumor indications specified in the National Medical Products Administration (NMPA )approved drug directions within 1 week before the first drug use;
  3. Imaging (Computed Tomography or Magnetic Resonance Imaging) shows that the tumor has invaded important blood vessels, or the researcher has determined that the tumor is highly likely to invade important blood vessels and cause fatal massive bleeding during subsequent studies;
  4. Uncontrolled pleural effusion, pericardial effusion, or moderate to severe ascites that still require repeated drainage;
  5. Known to have spinal cord compression, meningeal metastasis/malignant meningitis, accompanied by symptoms of brain metastasis, or symptoms/imaging control time less than 4 weeks. Within 2 weeks before the start of treatment, steroid therapy or dehydration agents are still required;
  6. For non-small cell lung cancer subjects known to have meaningful gene mutations such as epidermal growth factor receptor (EGFR) mutations, anaplastic lymphoma kinase (ALK) fusion, ROS Proto-Oncogene 1, Receptor Tyrosine Kinase (ROS) fusion, etc., they should have received corresponding targeted therapy;
  7. Subjects with known human epidermal growth factor receptor 2 (HER2) positive gastric/gastroesophageal junction cancer and breast cancer should have received corresponding anti HER2 treatment;
* Known to be allergic to research drug excipient components
* Previously received targeted FGFR2b monoclonal antibod therapy
* Previously received chemotherapy drugs used in the protocol (limited to subjects receiving combination therapy during the dose escalation phase only)
* Individuals who have participated in and used other anti-tumor clinical trial drugs within 4 weeks prior to their first medication.
* According to the judgment of the researchers, there are situations that seriously endanger the safety of the subjects or affect their ability to complete the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | During the first cycle. Each cycle is 28 days
  DLT will be defined as toxicities that meet pre-defined severity criteria(according to the NCI CTCAE v5.0 toxicity assessment criteria), and assessed as having a suspected relationship to study drug that occurred within the first cycle(28 days) of treatment.
Maximum tolerated dose (MTD) | During the first cycle. Each cycle is 28 days
  MTD was defined as the highest dose at which dose-limiting toxicity (DLT) occurred in less than 33% of patients.
Recommended Phase II Dose | During the first cycle. Each cycle is 28 days
  The recommended dosage for subsequent Phase II studies will be based on MTD (Maximum Tolerant Dose), pharmacokinetics, preliminary efficacy and safety comprehensively determined.
Objective Response Rate (ORR) (dose expansion phase) | Up to 2 years
  Defined as the percentage of Complete Response (CR) plus partial response (PR) assessed by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 criteria.

SECONDARY OUTCOMES:
Adverse event rate | Up to 2 years
  The occurrence of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs) evaluated by Common Terminology Criteria for Adverse Events (CTCAE) 5.0.
Objective Response Rate (ORR) (dose escalation phase) | Up to 2 years
  Defined as the percentage of Complete Response (CR) plus partial response (PR) assessed by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 criteria.
Disease control rate (DCR) | Up to 2 years
  Defined as the proportion of subjects with CR, PR, or Stable Disease (SD).
Duration of Response (DOR) | Up to 2 years
  Defined as the time from first documented response to documented disease progression.
Progress Free Survival (PFS) | Up to 2 years
  Defined as the time from the first dose of TQB2210 to the first occurrence of disease progression or death from any cause.
Overall Survival (OS) | Up to 2 years
  Overall survival refers to the time from the first treatment to death from any cause.
Pharmacokinetics: The area under the curve (AUC) | 2 hours pre-dose, 0,2,6,24,48,72,120,168 hours after dose on cycle1 day1 and cycle3 day1; 2 hours pre-dose on cycle1 day15 and cycle3 day15, each cycle is 28 days.
  The area under the curve (AUC) of serum concentration of TQB2210.
Pharmacokinetics:Peak concentration (Cmax) | 2 hours pre-dose, 0,2,6,24,48,72,120,168 hours after dose on cycle1 day1 and cycle3 day1; 2 hours pre-dose on cycle1 day15 and cycle3 day15, each cycle is 28 days.
  Maximum observed concentration (Cmax) of TQB2210 antibody.
Pharmacokinetics: T1/2 | 2 hours pre-dose, 0,2,6,24,48,72,120,168 hours after dose on cycle1 day1 and cycle3 day1; 2 hours pre-dose on cycle1 day15 and cycle3 day15, each cycle is 28 days.
  Terminal half-life (T1/2)
Pharmacokinetics: Apparent Clearance (CL/F) | 2 hours pre-dose, 0,2,6,24,48,72,120,168 hours after dose on cycle1 day1 and cycle3 day1; 2 hours pre-dose on cycle1 day15 and cycle3 day15, each cycle is 28 days.
  Apparent Clearance： Apparent clearance refers to the rate of drug removal in the body, which reflects the degree of drug elimination in the body, as well as the bioavailability of the drug in the body
Pharmacokinetics: Vss/F | 2 hours pre-dose, 0,2,6,24,48,72,120,168 hours after dose on cycle1 day1 and cycle3 day1; 2 hours pre-dose on cycle1 day15 and cycle3 day15, each cycle is 28 days.
  When the drug distribution in plasma and tissue reaches equilibrium, the drug distribution in the body body according to the plasma drug concentration at this time is the required body fluid volume called apparent distribution volume.
Immunogenicity: The incidence of drug-resistant antibodies (ADA) and neutralizing antibodies (NAb) | Cycle1 Day1, Cycle2 Day1, Cycle6 Day1; Cycle12 Day1: pre-dose 120 minutes; At the end of treatment visit (EOT) 30 days after the end of the infusion. Each cycle is 28 days.
  The incidence of drug-resistant antibodies (ADA) and neutralizing antibodies (NAb)

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Cancer Hospital of Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - ZhuJiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Provincial People's Hospital (The First Affiliated Hospital of Hunan Normal University), Changsha, Hunan
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang